CLINICAL TRIAL: NCT05650632
Title: A Multicenter, Phase 1b, Open-label Study to Evaluate Dose Optimization Measures and Safety of Etentamig (ABBV-383) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Assess Adverse Events of Intravenously (IV) Infused Etentamig (ABBV-383) in Adult Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-108; 2023-504674-38-00 (Other: EU CT)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; ABBV-383; B-Cell Maturation Antigen
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm A (Part 1): ABBV-383 Dose Escalation (Experimental): B-cell maturation antigen (BCMA) naïve participants will receive different doses of ABBV-383 in 28 day cycles.
  Interventions: Drug: Etentamig (ABBV-383)
- Arm A (Part 2): ABBV-383 Dose Expansion (Experimental): BCMA naïve participants will receive the dose of ABBV-383 dose A in 28 day cycles.
  Interventions: Drug: Etentamig (ABBV-383)
- Arm B: ABBV-383 BCMA Exposed (Experimental): Participants previously exposed to BCMA-targeted agents will receive ABBV-383 Dose A in 28 day cycles.
  Interventions: Drug: Etentamig (ABBV-383)
- Arm C: ABBV-383 Step Up (Experimental): Participants will receive step up dose and full target dose of ABBV-383 in 28 day cycles.
  Interventions: Drug: Etentamig (ABBV-383)
- Arm D: ABBV-383 Step Up (Experimental): Participants who have received at least 1 and no more than 3 prior lines of therapy will receive step up dose and full target dose of ABBV-383 in 28 day cycles.
  Interventions: Drug: Etentamig (ABBV-383)

INTERVENTIONS:
Drug: Etentamig (ABBV-383) — Intravenous Infusion

SUMMARY:
Multiple Myeloma (MM) is a cancer of the blood's plasma cells ( blood cell). The cancer is typically found in the bones and bone marrow (the spongy tissue inside of the bones) and can cause bone pain, fractures, infections, weaker bones, and kidney failure. Treatments are available, but MM can come back (relapsed) or may not get better (refractory) with treatment. This is a study to determine adverse events and change in disease symptoms of etentamig (ABBV-383) in adult participants with relapsed/refractory (R/R) MM.

Etentamig (ABBV-383) is an investigational drug being developed for the treatment of R/R Multiple Myeloma (MM). This study is broken into 4 Arms; Arm A (Parts 1 and 2), Arm B and Arms C & D. Arm A includes 2 parts: step-up dose optimization (Part 1) and dose expansion (Part 2). In Part 1, different level of step-up doses are tested followed by the target dose of etentamig (ABBV-383). In Part 2, the step-up dose identified in Part 1 (Dose A) will be used followed by the target dose A of etentamig (ABBV-383). In Arm B a flat dose of etentamig (ABBV-383) will be tested. In Arms C & D, the step-up dose identified in Arm A will be used followed by the target dose of etentamig (ABBV-383) to investigate outpatient administration of etentamig (ABBV-383). Around 210 adult participants with relapsed/refractory multiple myeloma will be enrolled at approximately 50 sites across the world.

Participants will receive etentamig (ABBV-383) as an infusion into the vein in 28 day cycles for approximately 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have measurable disease as outlined in the protocol.
* Eastern Cooperative Oncology Group (ECOG) performance of <= 2. Arm C and Arm D: ECOG performance of <= 1.
* Relapsed/refractory (R/R) multiple myeloma (MM) with documented evidence of progression during or after the participant's last treatment regimen based on the investigator's determination of the International Myeloma Working Group (IMWG) 2016 criteria.
* Must be naïve to treatment with etentamig (ABBV-383).
* Arm A: Must have received at least 3 or more lines of therapy, including a proteasome inhibitor (PI), an immunomodulatory imide drug (IMiD), and an anti-CD38 monoclonal antibody.
* Arm B: Must have received at least 2 or more lines of therapy, including exposure to a PI, an IMiD, an anti-CD38 monoclonal antibody, and a prior B-cell maturation antigen (BCMA)-targeted therapy (must be an anti-drug conjugate [ADC] or chimeric antigen receptor T-cell [CAR-T] directed against BCMA).
* Arm C: Must have received at least 2 or more lines of therapy, including exposure to a PI, an IMiD, and an anti-CD38 monoclonal antibody. Must be suitable for outpatient administration of etentamig (ABBV-383).
* Arm D: Must have received at least 1 and no more than 3 prior lines of therapy, including exposure to a PI, an IMiD, or an anti-CD38 monoclonal antibody. Must be suitable for outpatient administration of etentamig (ABBV-383).

Exclusion Criteria:

* Arm A: Received BCMA-targeted therapy.
* Arm C and Arm D: Rapidly progressing disease per investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Arm A (Part 1 and Part 2) Arm C, and Arm D: Number of Grade >= 2 Cytokine Release Syndrome (CRS) Events | Up to Day 28
  CRS is defined by fever, hypoxia, and hypotension and graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines
Arm B: Number of Adverse Events (AEs) of Special Interest (CRS and Immune Effector Cell-associated Neurotoxicity Syndrome [ICANS]) | Up to Day 28
  AEs of special interest will be graded according to American Society for Transplantation and Cellular Therapy (ASTCT) 2019 guidelines. All other AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Arm A, Arm C. and Arm D: Number of Cytokine Release Syndrome (CRS) Events | Up to 3 Years
  CRS is defined by fever, hypoxia, and hypotension and graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (22):
  - Mayo Clinic Arizona /ID# 251405, Phoenix, Arizona
  - Highlands Oncology Group - Springdale /ID# 267742, Springdale, Arkansas
  - Rocky Mountain Cancer Centers - Aurora /ID# 268574, Aurora, Colorado
  - Medical Oncology Hematology Consultants /ID# 268560, Newark, Delaware
  - Hope And Healing Cancer Services /ID# 268536, Hinsdale, Illinois
  - Fort Wayne Medical Oncology And Hematology /ID# 268179, Fort Wayne, Indiana
  - Tulane University School of Medicine /ID# 251204, New Orleans, Louisiana
  - Mayo Clinic - Rochester /ID# 251164, Rochester, Minnesota
  - NHO Revive Research Institute, LLC /ID# 267869, Lincoln, Nebraska
  - Mt Sinai /ID# 251166, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 251167, New York, New York
  - University of North Carolina /ID# 251203, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 251165, Winston-Salem, North Carolina
  - University Of Cincinnati Medical Center /ID# 251746, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center /ID# 267088, Eugene, Oregon
  - Vanderbilt Ingram Cancer Center /ID# 252470, Nashville, Tennessee
  - Texas Oncology - Central/South Texas /ID# 268563, Austin, Texas
  - Oncology Consultants /ID# 268323, Houston, Texas
  - Texas Oncology - Northeast Texas /ID# 268877, Tyler, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 268559, Fairfax, Virginia
  - Fred Hutchinson Cancer Center. /ID# 267940, Seattle, Washington
  - Northwest Medical Specialties Tacoma /ID# 267117, Tacoma, Washington
- Canada (2):
  - Juravinski Cancer Centre /ID# 252053, Hamilton, Ontario
  - Ottawa Hospital Research Institute /ID# 252151, Ottawa, Ontario
- Denmark (2):
  - Odense University Hospital /ID# 251261, Odense, Region Syddanmark
  - Vejle Sygehus /ID# 251260, Vejle, Region Syddanmark
- France (6):
  - Institut Paoli-Calmettes /ID# 252100, Marseille, Bouches-du-Rhone
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 252101, Créteil, Paris
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 251196, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 251223, Pierre-Bénite, Rhone
  - CHU Poitiers - La miletrie /ID# 251219, Poitiers, Vienne
  - AP-HP - Hopital Saint-Antoine /ID# 252326, Paris
- Israel (4):
  - Hadassah Medical Center-Hebrew University /ID# 252079, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 251329, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 251573, Tel Aviv, Tel Aviv
  - Rabin Medical Center. /ID# 251330, Petah Tikva
- Spain (3):
  - Hospital Universitario Marques de Valdecilla /ID# 251528, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 251545, Majadahonda, Madrid
  - Hospital Universitario de Salamanca /ID# 251529, Salamanca
- United Kingdom (2):
  - University College London Hospital /ID# 251357, London, Greater London
  - The Christie Hospital /ID# 251774, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-108